CLINICAL TRIAL: NCT03594162
Title: Compassionate Use Administration of Autologous CAR T Cells Targeting the CD19 Antigen and Containing the Inducible Caspase 9 Safety Switch
Brief Title: Compassionate Use of CAR T Cells Targeting the CD19 Antigen and Containing the Inducible Caspase 9 Safety Switch
Status: No longer available | Type: Expanded Access
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Bellicum Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: LCCC 1830-ATL-COM
Record Dates: First submitted 2018-07-03; First posted 2018-07-20 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2020-01

CONDITIONS: Acute Lymphoblastic Leukemia; Immune System Diseases; Immunoproliferative Disorders
Keywords: CAR T cells; CD19; Leukemia; T Lymphocytes; AP1903
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Immune System Diseases; Immunoproliferative Disorders; Leukemia | interventions — AP 1903 reagent; Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: iC9-CAR19 cells — One of two dose levels will be given: 1 x 10^5 or 5 x 10^5
  Other Names: CAR.CD19 T cells
Drug: AP1903 — Subjects who develop grade 4 CRS or grade 3 CRS that is refractory to standard of care interventions will be given AP1903 at .4 mg/kg.
  Other Names: Rimiducid
Drug: Cyclophosphamide — 900 mg/m^2 IV over 1 hour on day 4 of lymphodepleting chemotherapy.
  Other Names: Neosar
Drug: Fludarabine — 25 mg/m^2/day IV over 30 minutes administered for 3 consecutive days.
  Other Names: Fludara

SUMMARY:
This protocol for compassionate use combines 2 different ways of fighting disease: antibodies and T cells. Both antibodies and T cells have been used to treat patients with cancers, and both have shown promise, but neither alone has been sufficient to cure most patients. This protocol combines both T cells and antibodies to create a more effective treatment. The investigational treatment is called autologous T lymphocyte chimeric antigen receptor cells targeted against the CD19 antigen (ATLCAR.CD19) administration.

Prior studies have shown that a new gene can be put into T cells and will increase their ability to recognize and kill cancer cells. The new gene that is put in the T cells in this study makes a piece of an antibody called anti-CD19. This antibody sticks to leukemia cells because they have a substance on the outside of the cells called CD19. For this protocol, the anti-CD19 antibody has been changed so that instead of floating free in the blood part of it is now joined to the T cells. When an antibody is joined to a T cell in this way it is called a chimeric receptor. These CD19 chimeric (combination) receptor-activated T cells seem to kill some of the tumor, but they do not last very long in the body and so their chances of fighting the cancer are unknown.

Preliminary results have shown that many subjects receiving this treatment have experienced unwanted side effects including cytokine release syndrome. In this protocol, to help reduce cytokine release syndrome symptoms, the ATLCAR.CD19 cells have a safety switch that when active, can cause the cells to become dormant. These modified ATLCAR.CD19 cells with the safety switch are referred to as iC9-CAR19 cells. If the patient experiences moderate to severe cytokine release syndrome as a result of being given iC9-CAR19 cells, the patient can be given a dose of a second study drug, AP1903, if standard interventions fail to alleviate the symptoms of cytokine release syndrome. AP1903 activates the iC9-CAR19 safety switch, reducing the number of the iC9-CAR19 cells in the blood.

The primary purpose of this protocol is to treat a single patient with a second dose of iC9-CAR19 T cells.

DETAILED DESCRIPTION:
Lymphodepleting Chemotherapy:

The patient will receive a lymphodepleting regimen of fludarabine 25 mg/m2/day administered IV over 30 min for three consecutive days and a single IV dose of cyclophosphamide 900 mg/m2 administered over 1 hr on the fourth day.

Administration of iC9-CAR19 T cells:

Post lymphodepletion, if the patient meets eligibility criteria for cellular therapy, then will receive iC9-CAR19 T cells within 2-14 days after completing the pre-conditioning chemotherapy regimen. We will administer iC9-CAR19 post lymphodepletion at one of the following doses based on the percentage of circulating lymphoblasts prior to lymphodepletion: (1) dose of 5 x 10^5 transduced cells/kg or (2) dose of 1 x 10^5 transduced cells/kg.

Duration of Therapy:

Therapy under this compassionate use protocol involves 1 infusion of iC9-CAR19 cells.

Duration of Follow-up:

The patient will be followed for up to 15 years for replication-competent retrovirus evaluation or until death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria- Lymphodepletion

The patient must fulfill all of the following inclusion criteria to participate in this compassionate use protocol:

* Written informed consent for use of compassionate use therapy signed by patient or legal guardian of a pediatric patient.
* Age 3 to 17 years of age for pediatric patient (weight must be ≥ 10 kg), ≥ 18 to 70 years of age for an adult patient at the time of consent.
* Relapsed or refractory precursor B cell ALL:

  * Second or greater bone marrow relapse OR
  * Any bone marrow relapse >100 days after allogeneic stem cell transplant OR
  * Primary refractory ALL defined as no complete response after 2 cycles of a standard of care chemotherapy regimen OR
  * For an adult patient: first bone marrow relapse with duration of first CR <1 year OR CR1 duration ≥1 year and refractory to ≥1 cycle of therapy for treatment of relapse
  * A patient with isolated non-CNS extramedullary disease will be eligible as long as the time-of-remission criteria above for bone marrow relapses or primary refractory ALL are met and the biopsy for extramedullary disease confirms CD19 expression
  * For a pediatric patient: first bone marrow or isolated non-CNS extramedullary relapse refractory to 1 cycle of standard therapy for relapsed ALL
  * While active CNS3 leukemia will be excluded, any patient with concurrent CNS3 disease and bone marrow relapse who has responded to CNS-directed therapy prior to enrollment will be allowed to participate. Intrathecal chemotherapy will be allowed to continue between lymphodepleting chemotherapy and cell infusion.
  * Patients with CNS2 disease and concurrent bone marrow relapse will be eligible. Intrathecal chemotherapy will be allowed to continue between lymphodepleting chemotherapy and cell infusion
* Patients with Ph+ ALL will be eligible if they have failed ≥ 2 ABL tyrosine kinase inhibitors. Patients with the T315I ABL kinase point mutation will be eligible if they have failed ponatinib-containing therapy, regardless of the number of prior ABL tyrosine kinase inhibitors.
* CD19 positivity of lymphoblasts confirmed by flow cytometry or IHC per institutional standards.
* Karnofsky score > 60% if ≥16 years old or Lansky performance score of greater than 60% if <16 years old (See Appendix A: Performance Status (Lansky and Karnofsky)).
* Life expectancy ≥ 12 weeks.
* Patients who have received prior therapy with murine antibodies must have documentation of absence of human anti-mouse antibodies (HAMA) prior to lymphodepletion on this study.
* Demonstrate adequate renal and hepatic function as defined in the table below; all screening labs to be obtained within 72 hrs prior to lymphodepletion.

  * Serum Creatinine: ≤ 1.5 x ULN
  * Bilirubin: ≤ 1.5 x upper limit of normal (ULN), unless attributed to Gilbert's Syndrome
  * Aspartate Aminotransferase (AST): ≤ 3.0 × ULN
  * Alanine aminotransferase (ALT): ≤ 3.0 × ULN
  * For pediatric patients, adequate renal function is defined below:

Age Maximum Serum Creatinine (mg/dL) Male Female 3 to <6 years ≤0.8 ≤0.8 6 to <10 years ≤1 ≤1 10 to <13 years ≤1.2 ≤1.2 13 to <16 years ≤1.5 ≤1.4 16 to <18 years ≤1.7 ≤1.4

* Females of childbearing potential must have a negative serum pregnancy test within 72 hours prior to lymphodepletion. NOTE: Females are considered of child bearing potential unless they are premenarchal, surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months
* Females and males of childbearing potential must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 3 months after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method. Female patients will inform their male partners that they must use the methods of birth control required by the protocol.
* Male patients with female partners must have had a prior vasectomy or agree to use an adequate method of contraception (i.e., double barrier method: condom plus spermicidal agent) starting with the first dose of study therapy through 3 months after the last dose of study therapy.
* As determined by the enrolling physician or protocol designee, ability of the patient to understand and comply with compassionate use protocol procedures.
* Patients currently receiving "maintenance" doses of chemotherapy are eligible and the need for intrathecal prophylaxis prior to lymphodepletion is left to the discretion of the investigator. Maintenance chemotherapy is defined as methotrexate ≤30 mg/m2/week, mercaptopurine ≤100 mg/m2/day and vincristine ≤ 2 mg/28 days. For patients who receive chemotherapy, including intrathecal chemotherapy, that does not fit this definition of maintenance chemotherapy, a two week washout between the last dose of standard of care chemotherapy and the beginning of lymphodepletion will be required.
* Patients must have leftover autologous transduced activated T-cells from the LCCC 1541-ATL clinical protocol that meet the Certificate of Analysis (CofA) acceptance criteria.

Exclusion Criteria- Lymphodepletion

Patients meeting any of the following criteria CANNOT participate in this compassionate use protocol:

* Patients with relapsed fulminant CD19+ ALL that is rapidly progressing.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use if the milk is collected while the mother is being treated on study).
* Has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.
* Patients must not have tumor in a location where enlargement could cause airway obstruction.
* Patients may not have an oxygen requirement as defined by pulse oximetry of < 90% on room air.
* Treatment with any investigational drug within 14 days (i.e., two weeks) prior to lymphodepletion or has received any tumor vaccines within the previous five weeks prior to lymphodepletion.
* Patients with the following known systemic viral infections will be excluded: active HIV, HTLV, HBV, HCV.
* Patients who are on treatment for other active uncontrolled infections (not referenced above) with resolution of signs/symptoms are not excluded. Non-influenza, non-RSV, isolated upper respiratory infections are not excluded. Other active uncontrolled infections will be excluded.
* Use of systemic corticosteroids at doses ≥10mg/day prednisone or its equivalent; those receiving <10mg/day may be enrolled at discretion of investigator. (Note: Corticosteroid use with doses at the discretion of the treating physician are allowed after procurement up to the beginning of lymphodepletion.). Physiologic replacement with hydrocortisone is allowed at 6-12 mg/m2/day, or equivalent.

Inclusion Criteria- iC9-CAR19 Cell Infusion

Subjects must fulfill all of the following inclusion criteria to participate in this compassionate use protocol:

* Females and males of childbearing potential must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 3 months after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method. Female patients will inform their male partners that they must use the methods of birth control required by the protocol.
* Male patients with female partners must have had a prior vasectomy or agree to use an adequate method of contraception (i.e., double barrier method: condom plus spermicidal agent) starting with the first dose of study therapy through 3 months after the last dose of study therapy.
* As determined by the enrolling physician or protocol designee, ability of the patient to understand and comply with compassionate use protocol procedures.

Exclusion Criteria- iC9-CAR19 Cell Infusion

Subjects meeting any of the following criteria CANNOT be enrolled in this study:

* Corticosteroid use is contraindicated following iC9-CAR19 infusion unless medically necessary e.g., to treat CRS).
* Severe systemic uncontrolled disease or toxicities that develop after lymphodepletion may prompt exclusion from cell infusion at the discretion of the investigator.

Ages: 3 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Foster, MD, Principal Investigator — Assistant Professor Hematology-Oncology
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States